CLINICAL TRIAL: NCT00795236
Title: Melatonin Studies in Young Blind Children and Adolescents
Brief Title: Melatonin Studies of Totally Blind Children
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unique provision in the American Recovery and Reinvestment Act prevented approval of second year no-cost-extension in which completion of analyses were planned.
Sponsor: Oregon Health and Science University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: eIRB 4664; 2R01HD042125-06 (NIH)
Record Dates: First submitted 2008-11-19; First posted 2008-11-21 (Estimated); Results first posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Sleep Disorder; Blindness
Keywords: melatonin
MeSH Terms: conditions — Sleep Wake Disorders; Blindness | interventions — Melatonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Observational (No Intervention): Observe to determine free-running versus entrained status.
- Melatonin (Experimental): Subjects with free-running rhythms will take melatonin.
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Melatonin — One 0.5 mg tablet of melatonin will be taken by subjects who are free-running and willing to enter the intervention phase of the study. These subjects will take melatonin until entrainment status is confirmed or throughout the duration of the study.
  Arms: Melatonin

SUMMARY:
The purpose of this study is to learn more about abnormal body rhythms in blind boys and girls that keep them from falling asleep at bed-time or cause them difficulty staying alert during the day. The investigators hope to learn if there are any differences between the body rhythms of girls and boys. The investigators also want to investigate whether age or puberty have an effect on body rhythms.

DETAILED DESCRIPTION:
Subjects will be asked to collect saliva samples in their home hourly throughout the daytime, approximately every 2 weeks. Subjects may be monitored for up to a year, after which they will be discontinued from the study. If subjects are found to be naturally entrained to the 24-hour day, they will be monitored longitudinally for changes. Subjects will be discontinued after their monitoring period is over or after an entrained status has been confirmed. While no specific time commitment is required, we hope most subjects will participant for 4 months - 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Totally blind
* Between 5-8 yrs or 17-20 yrs of age

Exclusion Criteria:

* Pregnancy
* Light perception
* Low melatonin production
* Taking melatonin
* Co-morbid medical disorders (such as seizure disorders)

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2009-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Lewy, MD, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The PI has retired from the institution. Sincere efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.
Groups:
- Melatonin: Subjects with free-running rhythms will take melatonin.
  Melatonin : One 0.5 mg tablet of melatonin will be taken by subjects who are free-running and willing to enter the intervention phase of the study. These subjects will take melatonin until entrainment status is confirmed or throughout the duration of the study.
Period: Overall Study
Arm/Group | Melatonin | Observational
Started | 0 | 0
Completed | 0 (Unable to consistently obtain saliva DLMO in subjects and thus couldn't measure circadian period) | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The PI has retired from the institution. Sincere efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Melatonin | Observational | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: To Test for a Proportional Gender Difference in Circadian Status (Free-running Versus Entrained) in Blind Children and in Adolescents, a Chi-square Test of Significance Will be Used for Each Age Group.
Time Frame: Approximately 1 year
Population: as for baseline characteristics
Arm/Group | Observational | Melatonin
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: To Test for a Proportional Difference in Circadian Status (Free-running Versus Entrained) Between Pre and Post- Pubertal Males in Blind Boys and Young Men, a Chi-square Test of Significance Will be Used for Each Age Group.
Time Frame: Approximately 1 year
Population: as for baseline characteristics
Arm/Group | Melatonin | Observational
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: To Determine the Efficacy of Melatonin Treatment in Entraining Blind Free-running Children and Young Adults, a Binomial Test Will be Used.
Time Frame: Approximately 1 year
Population: as for baseline characteristics
Arm/Group | Melatonin | Observational
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The PI has retired from the institution. Sincere efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.
Arm/Group | Melatonin | Observational
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Technical problems with measurement leading to unreliable or uninterpretable data; Consistently could not obtain a complete melatonin profile from participants' saliva samplings and thus could not determine melatonin onset.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes